CLINICAL TRIAL: NCT00180531
Title: Monitoring of Arrhythmias and Heart Rate Variability in Patients With Congestive Heart Failure Treated With the Cardiac Resynchronisation Pacemaker Renewal TR2
Brief Title: Monitoring of Arrhythmias and HRV in Patients With Heart Failure Treated With the CRT Pacemaker Renewal TR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Responsible Party: Elisabeth Mouton, Guidant France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mona Lisa v. 1.1 3/12/03
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Renewal TR2

SUMMARY:
The objective of this study is to evaluate the prevalence of sustained ventricular and supraventricular rhythm disorders in patients implanted with a CONTAK RENEWAL TR2 ventricular resynchronization therapy (CRT) device

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe chronic heart failure, defined by the presence of NYHA class III or IV symptoms, Intra/interventricular synchronization disorder evaluated by echocardiography and/or Doppler Tissue Imaging (DTI, Yu's method22), Ejection fraction (EF) ≤ 40 %, If previous history of myocardial infarction, MI must be > 60 days from the date of inclusion, Estimated life expectancy > 6 months in the case of concomitant disease, Age ≥ 18 years, Optimal drug treatment of chronic heart failure (according to SFC* recommendations).

Exclusion Criteria:

* Conventional indication for treatment by implantable defibrillator upon inclusion, Cardiac transplant envisaged within 6 months, Unexplained syncope, MI < 60 days before inclusion, Non compliance to drug treatment for chronic heart failure, Any coronary pathology which may be treated by revascularisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of ventricular arrhythmias
Occurrence of supraventricular arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: P. CHEVALIER, MD, Principal Investigator — Hôpital Louis Pradel, Lyon; S Boveda, MD, Principal Investigator — Clinique Pasteur
Locations (10):
- France (10):
  - CHG Albi, Albi
  - CHU Michalon, Grenoble
  - CH La Croix Rousse, Lyon
  - Hôpital Louis Pradel, Lyon
  - Nouvelle Clinique Nantaise, Nantes
  - CHU Nîmes, Nîmes
  - CHG Perigueux, Périgueux
  - Hôpital Pontchaillou, Rennes
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Pasteur, Toulouse

REFERENCES:
- [Derived] Boveda S, Marijon E, Jacob S, Defaye P, Winter JB, Bulava A, Gras D, Albenque JP, Combes N, Pavin D, Delarche N, Teubl A, Lambiez M, Chevalier P; Mona Lisa Study Group. Incidence and prognostic significance of sustained ventricular tachycardias in heart failure patients implanted with biventricular pacemakers without a back-up defibrillator: results from the prospective, multicentre, Mona Lisa cohort study. Eur Heart J. 2009 May;30(10):1237-44. doi: 10.1093/eurheartj/ehp071. Epub 2009 Mar 4. PMID 19264750